CLINICAL TRIAL: NCT00780468
Title: A Pilot Study to Evaluate a Revised Method of Assessing Food in a Commercial Weight Management Program Format
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: WW International Inc (Industry)
Responsible Party: Principal Investigator, Lynne Becker, Project Manager, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR#18523
Record Dates: First submitted 2008-10-23; First posted 2008-10-27 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Obesity; Overweight
Keywords: Weight loss; Diet; Obesity
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Existing diet plan
  Interventions: Behavioral: Existing diet plan
- 2 (Experimental): New diet plan
  Interventions: Behavioral: New diet plan

INTERVENTIONS:
Behavioral: Existing diet plan
  Arms: 1
Behavioral: New diet plan
  Arms: 2

SUMMARY:
This study will provide data on two systems for assigning point values to food choices in a diet plan. The primary purpose of this study is to compare the effectiveness of the two systems with regard to changes in body weight.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 25-65 years of age inclusive
* Body Mass Index (BMI) 27.0 -35.0 inclusive.
* Not currently taking a prescription medication for weight loss (e.g. orlistat (Xenical), sibutramine (Meridia), phentermine).
* Not currently taking any over-the-counter weight loss medications or supplement(s).
* Not currently enrolled in commercial weight loss program (e.g. Jenny Craig, Weight Watchers) or self-help group (e.g. TOPS, Overeaters Anonymous).
* Willing and able to commit to regular physical activity (e.g. walking) five days per week as required by study protocol.
* Willing to keep and turn in a daily log/compliance book at the times required by study protocol.
* Willingness and ability to make all scheduled appointments at MUSC as required by study protocol.
* Willingness to make weekly meetings at MUSC.

Exclusion Criteria:

* History of thyroid disease, but not taking medication, or medication dosage changed one or more times over last 6 months. History of thyroid disease and on a stable dose of prescription medication for 6 months or longer is acceptable.
* Diagnosed with Type I or Type II diabetes or glucose intolerance, or use of anti-diabetic medications
* History of a surgical procedure for weight loss at any time (e.g. gastroplasty, gastric by-pass, gastrectomy or partial gastrectomy, adjustable banding, gastric sleeve).
* History of major surgery within three months of enrollment.
* History of heart problems (e.g. angina, bypass surgery, MI, etc.) within three months prior to enrollment.
* Presence of implanted cardiac defibrillator or pacemaker.
* Uncontrolled hypertension/high blood pressure.
* Orthopedic limitations that would interfere with ability to engage in regular physical activity.
* Gastrointestinal disorders including chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, chronic diarrhea or active gallbladder disease.
* History or presence of cancer. Persons with successfully resected basal cell carcinoma of the skin may be enrolled if treatment completed more than 6 months prior to enrollment.
* History of clinically diagnosed eating disorders including anorexia nervosa or bulimia nervosa.
* Women who are pregnant, lactating , trying to become pregnant or unwilling to use an effective means of birth control.
* Participation in another clinical trial within 30 days prior to enrollment.
* Weight loss of more than 5 pounds for any reason over the 30 days prior to enrollment.
* Taking any psychotropic medicine known to influence weight or weight loss

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Change in bodyweight. | 12 weeks

SECONDARY OUTCOMES:
Changes in waist circumference, blood pressure, lipids, questionnaire measures | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M. O'Neil, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina Weight Management Center, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Milsom VA, Malcolm RJ, Johnson GC, Pechon SM, Gray KM, Miller-Kovach K, Rost SL, O'Neil PM. Changes in cardiovascular risk factors with participation in a 12-week weight loss trial using a commercial format. Eat Behav. 2014 Jan;15(1):68-71. doi: 10.1016/j.eatbeh.2013.10.004. Epub 2013 Oct 21. PMID 24411753
- [Derived] O'Neil PM, Theim KR, Boeka A, Johnson G, Miller-Kovach K. Changes in weight control behaviors and hedonic hunger during a 12-week commercial weight loss program. Eat Behav. 2012 Dec;13(4):354-60. doi: 10.1016/j.eatbeh.2012.06.002. Epub 2012 Jun 28. PMID 23121787